CLINICAL TRIAL: NCT04509557
Title: [177Lu]Ludotadipep Treatment in Patients With Metastatic Castration-resistant Prostate Cancer: Phase I Clinical Trial.
Brief Title: [177Lu]Ludotadipep Treatment in Patients With Metastatic Castration-resistant Prostate Cancer.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: FutureChem (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: FC705-1
Record Dates: First submitted 2020-07-07; First posted 2020-08-12 (Actual); Last update posted 2022-10-20 (Actual); Status verified 2022-10

CONDITIONS: Metastatic Castration-resistant Prostate Cancer
Keywords: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Intervention Model Description: Dose is administered by differentiated into 5 groups (6 subjects each) and sequentially elevated starting from a low dose to a high dose (50±5 mCi, 75±8 mCi, 100±10 mCi, 125±13 mCi, 150±15 mCi).
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- 50mCi (Experimental): Using a drug product for which dose is determined (50±5 mCi dose), dilute with 0.9% NaCl 5 mL and slowly i.v. inject over 10 minutes, with 500 mL of 0.9% NaCl slowly administered for hydration over approximately 90 minutes from 30 minutes before treatment to 60 minutes after treatment.
  Interventions: Drug: [177Lu]Ludotadipep
- 75mCi (Experimental): Using a drug product for which dose is determined (75±8 mCi dose), dilute with 0.9% NaCl 5 mL and slowly i.v. inject over 10 minutes, with 500 mL of 0.9% NaCl slowly administered for hydration over approximately 90 minutes from 30 minutes before treatment to 60 minutes after treatment.
  Interventions: Drug: [177Lu]Ludotadipep
- 100mCi (Experimental): Using a drug product for which dose is determined (100±10 mCi dose), dilute with 0.9% NaCl 5 mL and slowly i.v. inject over 10 minutes, with 500 mL of 0.9% NaCl slowly administered for hydration over approximately 90 minutes from 30 minutes before treatment to 60 minutes after treatment.
  Interventions: Drug: [177Lu]Ludotadipep
- 125mCi (Experimental): Using a drug product for which dose is determined (125±13 mCi dose), dilute with 0.9% NaCl 5 mL and slowly i.v. inject over 10 minutes, with 500 mL of 0.9% NaCl slowly administered for hydration over approximately 90 minutes from 30 minutes before treatment to 60 minutes after treatment.
  Interventions: Drug: [177Lu]Ludotadipep
- 150mCi (Experimental): Using a drug product for which dose is determined (150±15 mCi dose), dilute with 0.9% NaCl 5 mL and slowly i.v. inject over 10 minutes, with 500 mL of 0.9% NaCl slowly administered for hydration over approximately 90 minutes from 30 minutes before treatment to 60 minutes after treatment.
  Interventions: Drug: [177Lu]Ludotadipep

INTERVENTIONS:
Drug: [177Lu]Ludotadipep — Dose is sequentially elevated starting from a low dose to a high dose (50±5 mCi, 75±8 mCi, 100±10 mCi, 125±13 mCi, 150±15 mCi). If DLT is observed in 2 or less of 6 subjects at each level, advance to the next step. If DLT is observed in 3 or more participants, no further subject will participate in the study at the relevant dose. Appropriateness of the dose elevation is evaluated 8-9 weeks after drug administration.

SUMMARY:
The study aims to evaluate the stability and efficacy after administration of [177Lu]Ludotadipep in patients with metastatic castration resistant prostate cancer (mCRPC), with dose-escalation applied to determine the appropriate dose.

DETAILED DESCRIPTION:
[18F]PSMA PET/CT is conducted at the 2nd screening and only PSMA PET/CT positive patients can be enrolled (PSMA RADS 4 or more).

Dose is administered by differentiated into 5 groups (6 subjects each) and sequentially elevated starting from a low dose to a high dose (50±5 mCi, 75±8 mCi, 100±10 mCi, 125±13 mCi, 150±15 mCi).

ELIGIBILITY:
Inclusion Criteria:

1. Among prostate cancer patients with blood testosterone ≤50ng/dL, mCRPC patients showing radiological progression after standard taxene-based anticancer treatment and 2nd generation hormone agent (abiraterone, enzalutamed, or both)) treatment or patients who are not eligible for such standard medical treatment at the discretion of an investigator or patients who refuse such standard treatment
2. Patients who are positive on the [18F]PSMA PET/CT imaging
3. Subjects who were fully informed by an investigator of the study objectives, details, and characteristics of the study drug prior to study enrollment, and had an informed consent form signed by the subject or caretaker or legally acceptable representative
4. Male patients aged 20 years or older
5. Subjects who are sexually active and have a female partner of childbearing potential should meet the followings

   * Subjects should consent to practice contraception by continuously using a male condom from screening, throughout the study, and for at least 6 months after the last dose of the study drug
   * Subjects should never donate sperms from screening, throughout the study, and for at least 6 months after the last dose of the study drug
   * Subjects with a partner who is a woman of childbearing potential (including a pregnant or breastfeeding mother) should consent to maintain sexual abstinence or practice double contraception throughout the study * Double contraception: Corresponding to 2 or more of the followings - use of a condom, use of a non-hormonal intrauterine device, use of a diaphragm, use of a cervical cap, a sexual partner who has been vasectomized at least 3 months (as of the first screening visit) or a sexual partner medically diagnosed to be sterile
6. ECOG _ Performance score ≤2
7. Life expectancy ≥6 months

Exclusion Criteria:

1. Subjects determined by an investigator to have a serious medical condition making study conduct difficult
2. Subjects corresponding to the following conditions 1) Glomerular filtration rate ≤40 ml/min, 2) hemoglobin level ≤10.0 g/dL, 3) white cell count ≤4.0 × 109/L, 4) platelet count ≤100 × 109/L, 5) total bilirubin level ≥1.5 x upper normal limit, 6) serum albumin level ≤3.0 g/dL, 7) active ischemic heart disease or heart failure (New York Heart Association Classification III-IV), 8) uncontrolled diabetes/hypertension, 9) hyperkalemia >6.0 mmol/L
3. Vulnerable subjects (the investigator involved in the study or his/her family, research staff or students of the investigator involved in the study)
4. Patients with a persistent malignancy other than the prostate cancer
5. Patients who participated in a therapeutic clinical trial within the past 30 days and administered an investigational product other than standard treatment
6. Patients are excluded if treatment other than the treatment provided in this study is determined more appropriate as determined by the investigator based on the patient and disease characteristics

Min Age: 20 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Male patients aged 20 years or older.
Enrollment: 30 (Actual)
Dates: Start 2020-10-14 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-06-30 (Actual)

PRIMARY OUTCOMES:
Dose-limiting toxicity | From date of randomization (IP administration (0h, visit3, Day 0 ~ 3)) until the date of grade 4 neutropenia, grade 3 febrile neutropenia, other grade 3 or 4 non-hematological toxicity resulting from [177Lu]Ludotadipep, persisting for 5 days or more.
  Dose-limiting toxicity is defined as CTCAE grade 4 thrombocytopenia (platelet count <25x109/L), grade 4 neutropenia (absolute neutrophil count (ANC) < 0.5 x 109), grade 3 febrile neutropenia (ANC <1000/mm3 and temperature >38.3℃ on at least 1 occasion or temperature ≥38℃ persisting for 1 hr), and other grade 3 or 4 non-hematological toxicity resulting from [177Lu]Ludotadipep, persisting for 5 days or more.

SECONDARY OUTCOMES:
PSA level assessment | screening(Day -31 ~ -20), , visit4 (Day10), visit5 (Day17), visit6(Day24), visit7(Day31), visit8(Day45), visit9(Day59), visit10 (Day87)
  Comparative assessment of the PSA level before and after administration of [177Lu]Ludotadipep
Radiological assessment | 2nd screeing(Day -19 ~ -1 ), visit7(Day31), visit9(Day59)
  Comparative assessment of the locations and the quantitative change of a lesion on [18F]PSMA PET/CT before and after administration of [177Lu]Ludotadipep, and assessment of the treatment response by comparing the intake of the target lesion from an imaging test at each time point.
Biodistribution | 2 hours, 24 hours (1 day), 48 hours (2 days), 72 hours (3 days) at visit3 (Day 0~3), visit 4(Day10)
  Assessment of the absorption (uptake) into the blood, lungs, liver, spleen, pancreas, kidneys, muscle, stomach, and tumor based on the level obtained from SPECT/CT imaging at 2 hours, 24 hours (1 day), 48 hours (2 days), 72 hours (3 days) and additionally perform planar scan at visit 4.
Whole-body absorbed dose | 2 hours, 24 hours (1 day), 48 hours (2 days), 72 hours (3 days) at visit3(Day 0~3)
  Calculation of the whole-body absorbed dose by evaluating the absorbed dose into the adrenals, brain, gallbladder, intestine, stomach, heart, kidney, liver, muscle, lungs, pancreas, red marrow, skin, spleen, testes, thymus, thyroid, and urinary bladder.
Safety assessment by baseline symptoms | Screening(Day -31 ~ -20), 2nd screening(Day -19 ~ -1)
  Assessment of adverse events occured from screening (Day -31) and 2nd screening(Day -31 ~ -20) before IP administration.
Safety assessment by adverse events | visit 3(Day 0 ~3), visit4 (Day10), visit5 (Day17), visit6(Day24), visit7(Day31), visit8(Day45), visit9(Day59), visit10 (Day87)
  Assessment of adverse events occured from IP administration (visit 3,Day 0~3) until visit10 (Day87)
Number of participants with abnormal signs and symptom as assessed through physical examination | Screening(Day -31 ~ -20), 2nd screening(Day -19 ~ -1), visit 3(Day 0~3), visit4 (Day 10), visit5 (Day 17), visit6(Day24), visit7(Day31), visit8(Day45), visit9(Day59), visit10 (Day87)
  Number of participants with abnormal signs and symptom as assessed through physical examination from screening(Day -31 ~ -20) to visit10 (Day87)
Systolic and diastolic blood pressure (mm Hg) | Screening(Day -31 ~ -20), 2nd screening(Day -19 ~ -1), visit 3(Day 0~3), visit4 (Day10), visit5 (Day17), visit6(Day24), visit7(Day31), visit8(Day45), visit9(Day59), visit10 (Day87)
  Assessment of masured value using systolic and diastolic blood pressure (mm Hg) from screening(Day -31 ~ -20) to visit10 (Day87)
Body temperature (degrees Celsius) | Screening(Day -31 ~ -20), 2nd screening(Day -19 ~ -1), visit 3(Day 0~3), visit4 (Day10), visit5 (Day17), visit6(Day24), visit7(Day31), visit8(Day45), visit9(Day59), visit10 (Day87)
  Assessment of masured value using body temperature (degrees Celsius) from screening(Day -31 ~ -20) to visit10 (Day87)
Pulse rate (beats per minute) | Screening(Day -31 ~ -20), 2nd screening(Day -19 ~ -1), visit 3(Day 0~3), visit4 (Day10), visit5 (Day17), visit6(Day24), visit7(Day31), visit8(Day45), visit9(Day59), visit10 (Day87)
  Assessment of masured value using pulse rate (beats per minute) from screening(Day -31 ~ -20) to visit10 (Day87)
Number of participants with abnormal hematology values | Screening(Day -31 ~ -20), visit 3(Day 0~3), visit4 (Day10), visit5 (Day17), visit6(Day24), visit7(Day31), visit8(Day45), visit9(Day59), visit10 (Day87)
  Number of participants with abnormal hematology values ( WBC, WBC differential, Hemoglobin, Hematocrit, RBC, Platelet, free lutetium -at 3 minutes, 15 minutes, 30 minutes, 60 minutes, 180 minutes, 24 hours, 48 hours, and 72 hours after IP administration) from screening(Day -31 ~ -20) to visit10 (Day87) except 2nd screening(Day -19 ~ -1).
Number of participants with abnormal chemistry values | Screening(Day -31 ~ -20), visit 3(Day 0~3), visit4 (Day10), visit5 (Day17), visit6(Day24), visit7(Day31), visit8(Day45), visit9(Day59), visit10 (Day87)
  Assessment of masured value using chemistry( free PSA, glucose, Total bilirubin, AST/ALT, Alkaline phosphatase, BUN/ Creatinine, Sodium, Potassium, Chloride, CA, Phosphorus, Total Protein, Albumin) from screening(Day -31 ~ -20) to visit10 (Day87) except 2nd screening(Day -19 ~ -1).
Number of participants with abnormal urinalysis values | Screening(Day -31 ~ -20), visit 3(Day 0~3), visit4 (Day10), visit5 (Day17), visit6(Day24), visit7(Day31), visit8(Day45), visit9(Day59), visit10 (Day87)
  Assessment of masured value using urinalysis (Specific Gravity, Protein, pH, Glucose, Occult Blood, Ketone) from screening(Day -31 ~ -20) to visit10 (Day87) except 2nd screening(Day -19 ~ -1).

CONTACTS AND LOCATIONS:
Overall Officials: Ji Youl Lee, Principal Investigator — The Catholic University of Korea
Locations (1):
- The Catholic University of Korea, Seoul, St, Mary's Hospital, 222, Banpo-daero, Seocho-gu, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Zhou J, Neale JH, Pomper MG, Kozikowski AP. NAAG peptidase inhibitors and their potential for diagnosis and therapy. Nat Rev Drug Discov. 2005 Dec;4(12):1015-26. doi: 10.1038/nrd1903. PMID 16341066
- [Background] Mease RC, Foss CA, Pomper MG. PET imaging in prostate cancer: focus on prostate-specific membrane antigen. Curr Top Med Chem. 2013;13(8):951-62. doi: 10.2174/1568026611313080008. PMID 23590171
- [Background] Lutje S, Heskamp S, Cornelissen AS, Poeppel TD, van den Broek SA, Rosenbaum-Krumme S, Bockisch A, Gotthardt M, Rijpkema M, Boerman OC. PSMA Ligands for Radionuclide Imaging and Therapy of Prostate Cancer: Clinical Status. Theranostics. 2015 Oct 18;5(12):1388-401. doi: 10.7150/thno.13348. eCollection 2015. PMID 26681984
- [Background] Maurer T, Eiber M, Schwaiger M, Gschwend JE. Current use of PSMA-PET in prostate cancer management. Nat Rev Urol. 2016 Apr;13(4):226-35. doi: 10.1038/nrurol.2016.26. Epub 2016 Feb 23. PMID 26902337
- [Background] Haberkorn U, Eder M, Kopka K, Babich JW, Eisenhut M. New Strategies in Prostate Cancer: Prostate-Specific Membrane Antigen (PSMA) Ligands for Diagnosis and Therapy. Clin Cancer Res. 2016 Jan 1;22(1):9-15. doi: 10.1158/1078-0432.CCR-15-0820. PMID 26728408